CLINICAL TRIAL: NCT07221474
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of V940 in Combination With Pembrolizumab and Chemotherapy as First-Line Treatment for Participants With Metastatic Squamous NSCLC (INTerpath-013)
Brief Title: A Study of V940/Placebo + Pembrolizumab and Chemotherapy in Metastatic Squamous Non-Small Cell Lung Cancer (V940-013)
Acronym: INTerpath-13
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V940-013; V940-013 (Other: MSD); U1111-1318-2495 (Registry Identifier: UTN); 2025-520902-37-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — pembrolizumab; Carboplatin; Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V940 + Pembrolizumab + Chemo (Experimental): Induction phase: Participants receive pembrolizumab 400 mg intravenous (IV) infusion on Day 1 of a six week cycle plus a platinum doublet chemotherapy regimen (carboplatin area under the curve (AUC) 6 mg/mL/min IV infusion every 3 weeks (Q3W) × 2 doses combined with either paclitaxel 200 mg/m^2 IV infusion Q3W × 2 doses OR nab paclitaxel 100 mg/m^2 IV infusion weekly × 6 doses). V940 1 mg intramuscular (IM) injection is administered on Days 1 and 22 of Cycle 2 Induction (Q3W) for up to 2 doses.
  Maintenance phase: Participants receive pembrolizumab 400 mg IV infusion on Day 1 every 6 weeks (Q6W) for up to 15 doses. V940 1 mg IM injection is administered on Days 1 and 22 (Q3W) for up to 7 doses during maintenance.
  Interventions: Biological: V940; Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel
- Placebo + Pembrolizumab + Chemo (Experimental): Induction phase: Participants receive pembrolizumab 400 mg intravenous (IV) infusion on Day 1 of a six week cycle plus a platinum doublet chemotherapy regimen (carboplatin area under the curve (AUC) 6 mg/mL/min IV infusion every 3 weeks (Q3W) × 2 doses combined with either paclitaxel 200 mg/m^2 IV infusion Q3W × 2 doses OR nab paclitaxel 100 mg/m^2 IV infusion weekly × 6 doses). Placebo intramuscular (IM) injection is administered on Days 1 and 22 of Cycle 2 Induction (Q3W) for up to 2 doses.
  Maintenance phase: Participants receive pembrolizumab 400 mg IV infusion on Day 1 every 6 weeks (Q6W) for up to 15 doses. Placebo IM injection is administered on Days 1 and 22 (Q3W) for up to 7 doses during maintenance.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Other: Placebo

INTERVENTIONS:
Biological: V940 — 1 mg Intramuscular (IM) Injection
  Other Names: mRNA-4157; Intismeran Autogene
  Arms: V940 + Pembrolizumab + Chemo
Biological: Pembrolizumab — 200 mg IV Infusion
  Other Names: MK-3475; KEYTRUDA®
Drug: Carboplatin — Area Under the Curve (AUC) 6 (mg/mL/min) IV Infusion
Drug: Paclitaxel — 200 mg/m^2 IV Infusion
Drug: Nab-paclitaxel — 100 mg/m^2 IV Infusion
Other: Placebo — Placebo matched to V940 IM injection
  Arms: Placebo + Pembrolizumab + Chemo

SUMMARY:
Researchers want to know if V940 (the study treatment) given with pembrolizumab and chemotherapy can treat metastatic treatment-naive squamous non-small cell lung cancer (NSCLC). V940 is designed to help a person's immune system attack their specific cancer.

The goal of this study is to learn if people who receive V940 with pembrolizumab and chemotherapy live longer overall and without the cancer growing or spreading compared to people who receive placebo with pembrolizumab and chemotherapy. A placebo looks like the study treatment but has no study treatment in it. Using a placebo helps researchers better understand the effects of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria include, but are not limited to:

* Has a histologically or cytologically confirmed diagnosis of squamous non-small cell lung cancer (NSCLC) (Stage IV: M1a, M1b, M1c1, M1c2, AJCC Staging Manual, Version 9). NOTE: Mixed tumors will be characterized by the predominant cell type; however, small cell elements are not permitted.
* Has measurable disease per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by the local site investigator/radiology
* Has provided a tissue sample that is collected either at the time of or after the diagnosis of metastatic disease AND is from a site not previously irradiated
* Adverse events (AEs) due to previous anticancer therapies must have recovered to ≤Grade 1. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤Grade 2 neuropathy are eligible
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy (ART)
* Hepatitis B surface antigen (HBsAg) positive participants are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load prior to randomization
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable. NOTE: Participants must have completed curative antiviral therapy at least 4 weeks prior to randomization
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 assessed within 7 days before randomization
* Has a life expectancy of at least 3 months
* Has adequate organ function

Exclusion Criteria:

Exclusion Criteria include, but are not limited to:

* Is HIV-infected with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has received prior treatment with a cancer vaccine, including another personalized cancer vaccine (PCV)
* Has received prior systemic anticancer therapy for their metastatic NSCLC
* Has received prior therapy with an anti-programmed cell death 1 protein (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), or anti-programmed cell death ligand 2 (anti-PD-L2) agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor. NOTE: Prior treatment with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent in the neoadjuvant or adjuvant setting for nonmetastatic NSCLC is allowed as long as therapy was completed at least 12 months before diagnosis of metastatic NSCLC
* Has received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids
* Has received radiation therapy to the lung that is >30 gray within 6 months of start of study intervention
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has severe hypersensitivity (≥Grade 3) to V940, pembrolizumab, or any of the protocol allowed chemotherapy agents and/or any of their excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has active infection requiring systemic therapy
* Has a history of stem cell/solid organ transplant
* Has not adequately recovered from major surgery or has ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2029-07-02 (Estimated); Study Completion 2031-05-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to ~32 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1). PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review (BICR) will be presented.
Overall Survival (OS) | Up to ~42 months
  OS, defined as the time from randomization to death due to any cause. OS will be presented.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to ~26 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience CR or PR as assessed by BICR will be presented.
Duration of Response (DOR) | Up to ~42 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Number of Participants who Experience an Adverse Event (AE) | Up to ~42 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who experience an AE will be presented.
Number of Participants who Discontinue Study Intervention Due to an AE | Up to ~24 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who discontinue study intervention due to an AE will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- Cleveland Clinic - Ohio ( Site 0016), Cleveland, Ohio, United States
- Argentina (2):
  - Instituto Alexander Fleming ( Site 0201), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Fundacion Estudios Clinicos ( Site 0207), Rosario, Santa Fe Province
- One Clinical Research ( Site 0402), Nedlands, Western Australia, Australia
- National Cheng Kung University Hospital ( Site 0601), Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/